CLINICAL TRIAL: NCT02112890
Title: Seroprevalence of Hepatitis A, Hepatitis B and Bordetella Pertussis in Mexico
Brief Title: Study to Assess Seroprevalence of Hepatitis A, Hepatitis B and Bordetella Pertussis in Mexico
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 201076
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Hepatitis A; Viral Hepatitis Vaccines
Keywords: Mexico; Adolescents; Hepatitis; Seroprevalence; Pertussis; Young adults
MeSH Terms: conditions — Hepatitis A; Hepatitis; Whooping Cough | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Stored serum samples of the selected subjects obtained from the ENSANUT 2012

GROUPS / COHORTS (1):
- Study Group: A random sample of subjects constituting adolescents and young adults (≥10 - ≤25 years of age) that participated in the ENSANUT 2012 in Mexico.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data of the selected subjects (through structured questionnaires and interviews) and stored serum samples obtained from the ENSANUT 2012. A subset database will be designed by the NIPH for the purpose of this study. Extracted data and laboratory results of the selected subjects will be captured in the study database.

SUMMARY:
This study will assess the seroprevalence of hepatitis A virus (HAV), hepatitis B virus (HBV) and Bordetella pertussis (B. pertussis) in adolescents and young adults in Mexico.

DETAILED DESCRIPTION:
A random sample of subjects constituting adolescents and young adults (≥10 - ≤25 years of age) will be selected from the total population that participated in the Encuesta Nacional de Salud y Nutrición (ENSANUT) 2012 in Mexico.

Data (through structured questionnaires and interviews) and stored serum samples of the selected subjects obtained from the ENSANUT 2012 will be used in this study. A subset database will be designed by the National Institute of Public Health (NIPH) for the purpose of this study. Extracted data and laboratory results of the selected subjects will be captured in this database.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for the ENSANUT 2012 was obtained according to local regulations from the subject/ from the parent(s)/ legally acceptable representative (LAR) of the subject.
* A male or female between and including 10 and 25 years of age, who previously participated in the ENSANUT 2012 in Mexico.

Exclusion Criteria:

* Information required for the study is not available or incomplete.
* Inadequate or insufficient serum sample to perform the laboratory tests for this study.
* Serum sample is wrongly identified.

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects constituting adolescents and young adults (≥10 - ≤25 years of age) from the total population that participated in the ENSANUT 2012 in Mexico.
Sampling Method: Probability Sample
Enrollment: 1603 (Actual)
Dates: Start 2014-12-10 (Actual); Primary Completion 2016-05-02 (Actual); Study Completion 2016-05-02 (Actual)

PRIMARY OUTCOMES:
Assessment of seropositivity status (defined as the percentage of subjects with antibody titres positive) for anti-HAV | During the study (approximately 12 months)
Assessment of seropositivity status (defined as the percentage of subjects with antibody titres positive) for anti-HBV (Hepatitis B core antibody [anti-HBc], Hepatitis B surface antigen [HBsAg]) and Hepatitis B surface antibody (anti-HBs) | During the study (approximately 12 months)
Assessment of seropositivity status (defined as the percentage of subjects with antibody titres positive) for Pertussis antibodies | During the study (approximately 12 months)

SECONDARY OUTCOMES:
Assesment of the difference in HAV, HBV and B. pertussis seropositivity rates among - Socioeconomic strata, - Regions, - Age groups, - Genders, - Risk groups, - Vaccination status for B. pertussis (if available) | During the study (approximately 12 months)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cuernavaca, Morelos, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for study 201076 can be found on the GSK Clinical Study Register — https://www.gsk-studyregister.com/study/5271